CLINICAL TRIAL: NCT07328737
Title: Efficacy and Safety of One vs Three Cycles of Hyperthermic Intraperitoneal Chemotherapy After Cytoreductive Surgery for Pseudomyxoma Peritonei: A Multicenter Randomized Controlled Study
Brief Title: One vs Three HIPEC Cycles After CRS for Pseudomyxoma Peritonei
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Yan Li, Professor of Oncology and Director of the Department of Peritoneal Oncology, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25814-4-02
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Pseudomyxoma Peritonei
MeSH Terms: conditions — Pseudomyxoma Peritonei

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Procedure: Three HIPEC sessions
- Control Group (Active Comparator)
  Interventions: Procedure: One HIPEC session

INTERVENTIONS:
Procedure: One HIPEC session — Receive only a single intraoperative HIPEC session following CRS.
  Arms: Control Group
Procedure: Three HIPEC sessions — Receive two additional HIPEC sessions after CRS+HIPEC (on post-operative day 2 and day 4) at reduced drug doses.
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of one versus three sessions of hyperthermic intraperitoneal chemotherapy (HIPEC) after cytoreductive surgery (CRS) for patients with pseudomyxoma peritonei (PMP).

The main questions it aims to answer are:

* Does receiving three HIPEC sessions lead to better Progression-Free Survival (PFS) and Overall Survival (OS) compared to one session?
* What are the differences in postoperative complications (e.g., infection, bowel obstruction, myelosuppression) and organ toxicity (e.g., liver/kidney injury) between the two regimens?
* How do the different treatment schedules impact patients' quality of life?

Researchers will compare the experimental group (3 HIPEC sessions) to the control group (1 HIPEC session) to investigate the efficacy and safety of the additional sessions.

Participants will:

* Be randomly assigned to one of two groups:

  1. Control Group: Receive only a single intraoperative HIPEC session following CRS.
  2. Experimental Group: Receive two additional HIPEC sessions after CRS+HIPEC (on post-operative day 2 and day 4) at reduced drug doses.
* Undergo scheduled safety checks for side effects on days 1, 3, 5, 7, and 10 post-HIPEC.
* Attend a follow-up visit at 1 month after CRS+HIPEC and, if eligible, receive 6 cycles of standard postoperative chemotherapy.
* Attend regular long-term follow-up visits for several years, which will include physical examinations, blood tests (for tumor markers), CT scans, and quality-of-life questionnaires (EORTC QLQ-C30 version 3.0).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consent to participate, sign informed consent, and be willing and able to comply with the study protocol;
2. Age 18-70 years;
3. Undergo CRS+HIPEC with pathological diagnosis of PMP of high grade with signet-ring cells, high grade, or low grade;
4. Karnofsky performance status (KPS) >60;
5. Adequate function of major organs as follows:

   1. Hematology: WBC ≥3.5×10^9/L, ANC ≥1.0×10^9/L, LC ≥0.5×10^9/L, PLT ≥80×10^9/L, Hb ≥90 g/L;
   2. Hepatic function: AST, ALT, and TBIL ≤2×upper limit of normal (ULN);
   3. Renal function: serum creatinine <1.2×ULN;
   4. Coagulation: APTT ≤1.5×ULN; INR or PT ≤1.5×ULN;
   5. Cardiopulmonary function sufficient to tolerate major surgery and HIPEC;

(5) Radiological Peritoneal Cancer Index (PCI) ≥15; (6) No local or systemic antitumor therapy within 1 month prior to CRS+HIPEC; (7) Adverse reactions from prior treatments have resolved before study initiation or, in the investigator's judgment, will not interfere with this study;

Exclusion Criteria:

1. Metastases to lung, brain, bone, or liver;
2. AST, ALT, or TBIL ≥2×ULN;
3. Serum creatinine ≥1.2×ULN;
4. Severe mesenteric contraction;
5. Major organ dysfunction that cannot support the planned procedures;
6. Concomitant hematological disorders or other malignancies;
7. Acute or subacute infectious disease;
8. History of allergy to cisplatin or docetaxel, or marked allergic diathesis or severe allergy history;
9. Psychiatric or psychological disorders preventing cooperation with treatment and efficacy evaluation;
10. Any other condition deemed unsuitable for enrollment by the investigator;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival rate | From randomization until 12 months postoperatively.
serious adverse events incidence | From randomization until 1 months postoperatively.

SECONDARY OUTCOMES:
progression-free survival | From randomization until 3 years postoperatively.
Overall survival | From randomization until 3 years postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Tsinghua University affiliated Beijing Tsinghua Changgung Hospital, Beijing, Changping, China

IPD SHARING:
Plan to Share IPD: Undecided